CLINICAL TRIAL: NCT06241066
Title: The Prognostic Value of Tertiary Lymphatic Structure in Esophageal Squamous Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: bc2023192
Record Dates: First submitted 2024-01-25; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-12

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Surgery alone group: Patients who were diagnosed with esophageal squamous cell carcinoma and underwent esophageal squamous cell carcinoma resection without any prior treatment are included in this group. These patients had not been diagnosed with any other cancer. Finally, 96 patients were included.
  Interventions: Other: no-Intervention
- Neoadjuvant chemotherapy group: Patients who were diagnosed with esophageal squamous cell carcinoma and underwent esophageal squamous cell carcinoma resection, and underwent routine chemotherapy before surgery were included in this group. These patients were not diagnosed with any other cancers Finally, 89 patients were included.
  Interventions: Other: no-Intervention
- Neoadjuvant chemotherapy combined with immunotherapy group: Patients who were diagnosed with esophageal squamous cell carcinoma and underwent esophageal squamous cell carcinoma resection, and underwent routine chemotherapy combined with immunotherapy before surgery were included in this group. These patients were not diagnosed with any other cancers Finally, 81 patients were included.
  Interventions: Other: no-Intervention
- Neoadjuvant chemotherapy combined with radiotherapy group: Patients who were diagnosed with esophageal squamous cell carcinoma and underwent esophageal squamous cell carcinoma resection, and underwent routine chemotherapy combined with radiotherapy before surgery were included in this group. These patients were not diagnosed with any other cancers Finally, 93 patients were included.
  Interventions: Other: no-Intervention

INTERVENTIONS:
Other: no-Intervention — no-Intervention

SUMMARY:
Retrospective analysis of the presence and maturity of tertiary lymphoid structures in pathological sections of patients with esophageal squamous cell carcinoma after surgical treatment. Pay attention to the overall survival and disease free survival of these esophageal squamous cell carcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Pathologically diagnosed as esophageal squamous cell carcinoma; 2. Surgery for esophageal cancer; 3. Complete medical records;

Exclusion Criteria:

* Patients with a previous history of malignant tumor

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients pathologically confirmed esophageal squamous cell carcinoma(ESCC) who underwent complete surgical resection at Tianjin Medical University Cancer Hospital between 2014 and 2021
Sampling Method: Non-Probability Sample
Enrollment: 359 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
OS | The time from treatment to death or last follow-up, assessed up to 100 months.
  Overall Survival
DFS | The time from treatment to the first recurrence or last follow-up, assessed up to 100 months.
  Disease-free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Wencheng Zhang, M.D., Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Cancer Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No